CLINICAL TRIAL: NCT01050114
Title: A Double-Blind, Randomized Study of the Safety and Efficacy of OnabotulinumtoxinA (OnaBoNT-A) Versus Oral Oxybutynin in Spinal Cord Injured Patients With Neurogenic Detrusor Overactivity (Protocol Number 11-09-10-04)
Brief Title: OnabotulinumtoxinA (onaBoNT-A) Versus Oral Oxybutynin ER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christopher Patrick Smith (Other)
Responsible Party: Sponsor-Investigator, Christopher Patrick Smith, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-09-10-04 (BCM H-26296); H-26296 (Other: Baylor College of Medicine)
Record Dates: First submitted 2010-01-11; First posted 2010-01-15 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Overactive Bladder
Keywords: Botulinum Toxin; Oxybutynin; Overactive Bladder; Spinal Cord Injury; Urinary Incontinence; Nerve Growth Factor; Urine Biomarkers
MeSH Terms: conditions — Urinary Bladder, Overactive; Spinal Cord Injuries; Urinary Incontinence; Hereditary Sensory and Autonomic Neuropathies | interventions — onabotulinum toxin A; Botulinum Toxins, Type A; Tolterodine Tartrate; oxybutynin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARM 1: onaBoNT-A injection + placebo (Other): onaBoNT-A 200 U (treatment 1)/ onaBoNT-A 200 U (treatment 2)/ onaBoNT-A 200 U (treatment 3) and placebo oral capsule daily
  Interventions: Drug: onaBoNT-A
- ARM 2: Placebo injection + oxybutynin ER (Other): Placebo injection (treatment 1)/ onaBoNT-A 200 U (treatment 2)/ onaBoNT-A 200 U (treatment 3) and oxybutynin ER 10 mg capsule daily
  Interventions: Drug: Oxybutynin ER

INTERVENTIONS:
Drug: onaBoNT-A — onaBoNT-A will be the active formulation. Each vial of onaBoNT-A Purified Neurotoxin Complex, Formulation No. 9060X, contains: 100 units (U) of Clostridium botulinum toxin type A, 0.5 mg albumin (human), and 0.9 mg sodium chloride in a sterile, vacuum-dried form without a preservative. One U corresponds to the calculated median lethal intraperitoneal dose (LD50) in mice. A 0.9% sterile saline (without preservative) for injection will be used as diluent for onaBoNT-A.
  Each treatment session will be administered as 20 injections each of 1 mL (10U/ml), evenly distributed into the bladder.
  Other Names: onabotulinumtoxinA; BOTOX(R)
  Arms: ARM 1: onaBoNT-A injection + placebo
Drug: Oxybutynin ER — Oxybutynin ER in a 10 mg capsule will be taken twice a day for the course of the study.
  Other Names: Ditropan XL; Urotrol; Oxytrol
  Arms: ARM 2: Placebo injection + oxybutynin ER

SUMMARY:
Overactive bladder is a condition associated with symptoms of feeling the urge to urinate, urinating often, and may or may not be accompanied by leakage of urine. A patient who has a spinal cord injury (SCI) often suffers from an overactive bladder which often leads to urinary incontinence (UI - an unwanted leakage of urine).

OnaBoNT-A bladder injections have been studied in clinical research trials. The results have shown an improvement in urinary symptoms by reducing how often urine leakage occurs and by increasing the amount of urine the bladder can hold.

This purpose of this clinical trial is to see if onaBoNT-A is safe and effective when injected into the bladder for the treatment of UI and if it works better than a drug that is taken by mouth. A second purpose of the study is to perform research tests on the urine samples provided by the volunteers. Urine presents a rich source of information for bladder diseases and the biomarkers (the chemical make-up of the urine cells) will be examined to learn if there are yet undiscovered reasons for urinary diseases. These tests would be very beneficial because the results would lead to better treatment of the urinary diseases.

Volunteers will be randomized to either: ARM 1: onaBoNT-A 200 U bladder injection and placebo oral capsule daily or ARM 2: Placebo bladder injection (saline) and oxybutynin ER 10mg capsule twice a day.

The treatments are onaBoNT-A bladder injection and a placebo oral capsule once a day or placebo bladder injection and oxybutynin ER (like Ditropan) capsule twice a day. Placebo contains no active medicine. Participation in this study will be about 6-7 months and involve 5 visits to the clinic. The risks of bladder onaBoNT-A

DETAILED DESCRIPTION:
Current treatment of neurogenic bladder dysfunction (NGB) is limited by the suboptimal results achieved using standard antimuscarinic agents. A prominent role for the actions of alternative transmitters/growth factors in peripheral micturition pathways is emerging from the growing number of pharmacologic and localization studies in humans. For example, recently published data demonstrates a significant increased expression of Nerve Growth Factor and chemokine/cytokine levels in patients with detrusor overactivity and NGB. Treatment with onabotulinumtoxinA (onaBoNT-A) not only was shown to reduce detrusor overactivity and improve urinary symptoms but also significantly reduced tissue and urine levels of factors such as NGF. Up to this point, no study has directly compared the effects of front-line therapy of antimuscarinic agents versus onaBoNT-A on urinary symptoms in patients with NGB resulting from spinal cord injury (SCI). In addition, no investigation has examined the effects that antimuscarinic agents or onaBoNT-A have on urinary levels of NGF and chemokines/cytokines, whether changes in urinary levels predict a clinical response or a return in symptoms, and if changes in urinary levels predate changes in clinical response.

Access to selective and reliable urine testing of NGF and chemokines/cytokines provides the unique opportunity to assess the impact that modulating these agents has on bladder function. The main purpose of this proposal is to incorporate novel urine biomarker testing into existing clinical methodologies in order to: 1) evaluate the safety and efficacy of 200 U onaBoNT-A injected into the detrusor versus oral oxybutynin for the treatment of urinary incontinence (UI) caused by neurogenic detrusor overactivity (NDO) in spinal cord injured patients and 2) to determine the potential role of urine biomarkers in guiding the process of patient selection and identify surrogate predictors of treatment outcomes.

This will be a double-blind, randomized, placebo-controlled, parallel-group study to assess the safety and efficacy of onaBoNT-A or 10 mg twice a day of oral oxybutynin hydrocholoride in spinal cord injured patients diagnosed with neurogenic detrusor overactivity.

Volunteers will include both males and females with spinal cord injuries who are 18 to 80 years of age.

Volunteers will be randomized using a blocked randomization approach to either:

ARM 1: onaBoNT-A 200 U bladder injection and placebo oral capsule daily or

ARM 2: Placebo bladder injection (saline) and oxybutynin ER 10mg capsule twice a day.

Subjects will be randomized into one of the two treatment arms, using a block size of 4. The order in which the treatments are assigned in each block is randomized and this process is repeated for consecutive blocks of subjects until all subjects are randomized. This process ensures that after every fourth randomized subject, the number of subjects in each treatment group is equal.

There will be five study visits over approximately 6-7 months.

The significance of these experiments begins with the fact that our proposed intervention is the first randomized clinical trial comparing the effects of onaBoNT-A (onabotulinumtoxinA) bladder injection versus anticholinergic medication for detrusor hyperreflexia (DH). In addition, this is the first study profiling urine levels of the signaling protein nerve growth factor (NGF) and chemokines/cytokines as possible bio-markers of bladder overactivity in patients with neurogenic detrusor overactivity. Finally, this is the only study to date comparing the effects that onaBoNT-A or anticholinergic medications have on urine NGF and chemokine/cytokine levels. If our hypotheses prove to be correct, the significance to treating patients with spinal cord injury with botulinum toxin A will be less incontinence, the requirement of lower doses or avoidance of anticholinergic medication and its associated side effects, and the ability to prevent the complications of DH/DESD (Detrusor-External Sphincter Dyssynergia) including urinary tract infections, decubiti, and impairment of quality of life. Although this study as written is of moderate length (i.e. total 4 years), we hope that by finding significant results, we will be able to capture a longitudinal history of this population by extending follow-up to a longer duration (i.e. over 10 years).

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 18 to 80 years old, weighing 110 pounds or more.
* urinary incontinence as a result of neurogenic detrusor overactivity for a period of at least 3 months prior to screening as a result of spinal cord injury
* must have a stable neurological injury occurring at least 6 months or more.
* has detrusor overactivity demonstrated during the screening period or within 1 year of screening.
* has a negative pregnancy result if female and of childbearing potential.

The following criteria are also required for entry into the study at Randomization/Day 1:

* experiences at least 14 episodes or more of urinary incontinence per week with no more than 2 incontinent-free days.
* currently uses or is willing to use clean intermittent catheterization (CIC) to empty the bladder (indwelling catheter is not permitted).
* Volunteers with a negative urine culture result must take an antibiotic medication for 3 days immediately prior to Randomization/Day 1 and agree to continue antibiotic medication for at least 3 days following treatment. Volunteers with a positive urine culture result indicating urinary tract infection (UTI), must take an antibiotic to which the identified organism is sensitive for at least 3 days immediately prior to Randomization/Day 1, on Randomization/Day 1, and continue for 3 days following the procedure (or longer as needed).

Exclusion Criteria:

* has history or evidence of any pelvic or urological abnormalities including but not limited to the following:

  1. elevated serum creatinine more than 2 times the upper limit of normal (reference range)
  2. current or history of hematuria, 1) if the hematuria is determined to be a pathologic condition or 2) is uninvestigated
  3. interstitial cystitis in the opinion of the investigator bladder stones within 6 months of screening
  4. surgery or bladder disease other than detrusor overactivity that may impact bladder function with the exception of surgeries for bladder stones (more than 6 months) and stress incontinence, uterine prolapse, rectocele, or cystocele (more than1year) from screening.
* has had previous or current botulinum toxin therapy within 9 months.
* has been immunized for any botulinum toxin serotype.
* discontinued anticholinergic medication for overactive bladder less than 14 days prior to Randomization/Day 1.
* has a history or current diagnosis of bladder cancer.
* male with previous or current diagnosis of prostate cancer or has a Prostate Specific Antigen (PSA) level greater than 10.0 ng/mL.
* has 24 hour total volume voided more than 3000 mL of urine
* has a post void residual volume above 200 mL.
* has an active genital infection, other than genital warts, either concurrently or within 4 weeks prior to screening.
* uses any anti-platelet or anticoagulant therapy or is using medications with anticoagulative effects within 3 days prior to treatment.
* has hemophilia or other clotting factor deficiencies or disorders that cause bleeding diatheses.
* has had concurrent treatment or treatment within 6 months of Randomization/Day 1 with capsaicin or resiniferatoxin.
* currently using or plans to use an implanted or non-implantable electrostimulation/ neuromodulation device for treatment of overactive bladder.
* has a known allergy or sensitivity to any components of the study medication, anesthetics or antibiotics or any other products associated with the treatment and general study procedures.
* has any medical condition that may put the volunteer at increased risk with exposure to onaBoNT-A including diagnosed myasthenia gravis, Eaton-Lambert syndrome or amyotrophic lateral sclerosis.
* female and pregnant, nursing or planning a pregnancy during the study, or of childbearing potential and unable or unwilling to use a reliable form of contraception during the study.
* currently or has previously participated in another therapeutic drug or device study within 30 days of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 12 weeks
  The primary endpoint is the reduction in mean weekly incontinent episodes in the onaBoNT-A treated group compared to the oxybutynin treated group at 12 weeks.

SECONDARY OUTCOMES:
The utility of urinary inflammatory markers as statistically significant predictors of treatment response. | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P. Smith, MD, Study Director — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - TIRR-Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Data will be published in aggregate.

REFERENCES:
- [Background] O'Leary M, Erickson JR, Smith CP, McDermott C, Horton J, Chancellor MB. Effect of controlled-release oxybutynin on neurogenic bladder function in spinal cord injury. J Spinal Cord Med. 2003 Summer;26(2):159-62. doi: 10.1080/10790268.2003.11753678. PMID 12828295
- [Background] Smith CP, Chancellor MB. Emerging role of botulinum toxin in the management of voiding dysfunction. J Urol. 2004 Jun;171(6 Pt 1):2128-37. doi: 10.1097/01.ju.0000127725.48479.89. PMID 15126771
- [Background] Smith CP, Nishiguchi J, O'Leary M, Yoshimura N, Chancellor MB. Single-institution experience in 110 patients with botulinum toxin A injection into bladder or urethra. Urology. 2005 Jan;65(1):37-41. doi: 10.1016/j.urology.2004.08.016. PMID 15667859
- [Background] Liu HT, Tyagi P, Chancellor MB, Kuo HC. Urinary nerve growth factor but not prostaglandin E2 increases in patients with interstitial cystitis/bladder pain syndrome and detrusor overactivity. BJU Int. 2010 Dec;106(11):1681-5. doi: 10.1111/j.1464-410X.2009.08851.x. PMID 19751258
- [Background] Tyagi P, Barclay D, Zamora R, Yoshimura N, Peters K, Vodovotz Y, Chancellor M. Urine cytokines suggest an inflammatory response in the overactive bladder: a pilot study. Int Urol Nephrol. 2010 Sep;42(3):629-35. doi: 10.1007/s11255-009-9647-5. Epub 2009 Sep 26. PMID 19784793